CLINICAL TRIAL: NCT04517318
Title: A Multi-center Study of the Treatment Patterns and Clinical Outcomes of Subsequent Therapies After Progression on Palbociclib in HR+/HER2- Metastatic Breast Cancer
Brief Title: Treatment After Palbociclib-containing Regimens
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-9
Record Dates: First submitted 2020-08-16; First posted 2020-08-18 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the prescription patterns and treatment outcomes of subsequent therapies after progression on palbociclib in the real world.

ELIGIBILITY:
Inclusion Criteria:

1. woman, age > 18 years old
2. Diagnosed with HR+/HER2- Metastatic Breast Cancer
3. Patients received at least one-cycle next-line treatment after progression on combined palbociclib and endocrine therapy
4. Complete medical history was available

Exclusion Criteria:

1. Medical history was incomplete

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer (according to International Classification of Diseases-10, ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression free survival
Adverse events | 6 weeks
  Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0)

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li Y, Li W, Gong C, Zheng Y, Ouyang Q, Xie N, Qu Q, Ge R, Wang B. A multicenter analysis of treatment patterns and clinical outcomes of subsequent therapies after progression on palbociclib in HR+/HER2- metastatic breast cancer. Ther Adv Med Oncol. 2021 Jun 11;13:17588359211022890. doi: 10.1177/17588359211022890. eCollection 2021. PMID 34178122